CLINICAL TRIAL: NCT01053793
Title: A Trial to Measure the Glycemic Index and Polyphenol Bioavailability of Four Different Varieties of Potato.
Brief Title: Glycemic Index and Polyphenol Bioavailability of Potatoes
Acronym: GI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guelph Food Research Centre (Other Government)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Dr. Dan Ramdath - Research Scientist, Agriculture and Agri-Food Canada - Guelph Food Research Centre
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 09-11-004; GFRC 09-11-004 (Other: Canadian Shield)
Record Dates: First submitted 2010-01-20; First posted 2010-01-21 (Estimated); Last update posted 2011-01-17 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes; Insulin Resistance
Keywords: Glycemic index; Anthocyanin; Potato; Polyphenol
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glucose Standard (Active Comparator)
  Interventions: Other: Glycemic response to different varieties of potatoes
- Potato Variety (Experimental)
  Interventions: Other: Glycemic response to different varieties of potatoes

INTERVENTIONS:
Other: Glycemic response to different varieties of potatoes — the glycemic response top 50g available carbohydrates from 4 potato varieties will be compared to a 50g glucose standard
  Other Names: Purple potato; Red potato; White potato; Yellow potaot

SUMMARY:
The purpose of this study is to determine the glycemic index of four varieties of potatoes and to determine the bioavailability of polyphenols contained in these potatoes.

DETAILED DESCRIPTION:
Ten healthy persons will have a fasting blood sample drawn and asked to randomly consume a 50g glucose drink (2 occasions), or 50g carbohydrate equivalent of cooked purple, red, yellow and white potatoes. Further blood samples will be obtained at 15,30, 45, 60, 90, 120, 180, 240 mins. Bloods from the first 2 hours will be analyzed for glucose and insulin to determine the glycemic response. Hourly blood samples will be analyzed for polyphenol to determine the bioavailability of polyphenols from the different potato variety. Urine samples will be collected before ingestion of the food items and again at 4 hours, and will be used to determine polyphenol bioavailability.

ELIGIBILITY:
Inclusion Criteria:

* healthy, non-smoker on no medication
* normal glucose tolerance
* willing to have a catheter inserted in forearm

Exclusion Criteria:

* abnormal glucose tolerance
* abnormal BMI
* on medication for a chronic disorder

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Glycemic response | 2 hrs

SECONDARY OUTCOMES:
Bioavailability of polyphenols from potatoes | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dan Ramdath, PhD, Principal Investigator — Agriculture and Agri-Food Canada; Maggie Laidlaw, PhD, Study Director — Nutracource Diagnostics Inc
Locations (1):
- Nutrasource Diagnostic Inc, Guelph, Ontario, Canada

REFERENCES:
- [Background] Wolever TM, Brand-Miller JC, Abernethy J, Astrup A, Atkinson F, Axelsen M, Bjorck I, Brighenti F, Brown R, Brynes A, Casiraghi MC, Cazaubiel M, Dahlqvist L, Delport E, Denyer GS, Erba D, Frost G, Granfeldt Y, Hampton S, Hart VA, Hatonen KA, Henry CJ, Hertzler S, Hull S, Jerling J, Johnston KL, Lightowler H, Mann N, Morgan L, Panlasigui LN, Pelkman C, Perry T, Pfeiffer AF, Pieters M, Ramdath DD, Ramsingh RT, Robert SD, Robinson C, Sarkkinen E, Scazzina F, Sison DC, Sloth B, Staniforth J, Tapola N, Valsta LM, Verkooijen I, Weickert MO, Weseler AR, Wilkie P, Zhang J. Measuring the glycemic index of foods: interlaboratory study. Am J Clin Nutr. 2008 Jan;87(1):247S-257S. doi: 10.1093/ajcn/87.1.247S. PMID 18175765
- [Background] Ramdath DD, Isaacs RL, Teelucksingh S, Wolever TM. Glycaemic index of selected staples commonly eaten in the Caribbean and the effects of boiling v. crushing. Br J Nutr. 2004 Jun;91(6):971-7. doi: 10.1079/bjn20041125. PMID 15182400
- [Background] Wolever TM, Vorster HH, Bjorck I, Brand-Miller J, Brighenti F, Mann JI, Ramdath DD, Granfeldt Y, Holt S, Perry TL, Venter C, Xiaomei Wu. Determination of the glycaemic index of foods: interlaboratory study. Eur J Clin Nutr. 2003 Mar;57(3):475-82. doi: 10.1038/sj.ejcn.1601551. PMID 12627186
- [Background] Wolever TM, Isaacs RL, Ramdath DD. Lower diet glycaemic index in African than South Asian men in Trinidad and Tobago. Int J Food Sci Nutr. 2002 Jul;53(4):297-303. doi: 10.1080/09637480220138142. PMID 12090025